CLINICAL TRIAL: NCT01436929
Title: Effect of Prophylactic Use of Silymarin on Hepatotoxicity Induced by Anti-tuberculosis Drugs
Acronym: PESOHHERZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRMH-06-2011-75; BRMH-06-2011-75 (Other: SeoulNUH)
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Tuberculosis
Keywords: silymarin; hepatotoxicity; tuberculosis; HREZ
MeSH Terms: conditions — Tuberculosis | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silymarin (Experimental): Silymarin: prophylactic administration of silymarin with anti-TB drugs Placebo: prophylactic administration of placebo with anti-TB drugs
  Interventions: Drug: Silymarin
- Placebo (Placebo Comparator): administration of placebo with anti-TB drugs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin — Silymarin 140mg 1tab bid for 8 weeks
  Arms: Silymarin
Drug: Placebo — Placebo 1tab bid
  Arms: Placebo

SUMMARY:
Tuberculosis is a worldwide common infectious disease and effective first line anti-tuberculosis (TB) drugs were available such as isoniazid, rifampicin, ethambutol, and pyrazinamide. However, anti-TB drugs may induce hepatic injury resulting in discontinuation of anti-TB drugs or changing anti-Tb drug regimen.

Silymarin has been widely studied for the effect on hepatitis and it has been used in hepatology.

Therefore, the investigators hypothesized that prophylactic administration of silymarin with anti-TB drugs may decrease the incidence and severity of hepatotoxicity induced by anti-TB drugs.

ELIGIBILITY:
Inclusion Criteria:

* subjects who are diagnosed with tuberculosis based on microbiological, biomolecular, pathological, or radiographical findings and are expecting to be administered with anti-tuberculosis drugs including INH, RFP, or PZA.
* adults >=35 years old

Exclusion Criteria:

* basal AST >40 IU/uL or ALT >40 IU/uL
* pregnancy
* lactating women
* cases with history of adverse events to silymarin

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
incidence of hepatotoxicity | 8 weeks
  the presence of hepatotoxicity will be evaluated at 2weeks, 4weeks, and 8weeks after initiation of anti-TB drugs. An interim analysis will be done after enrolling first 300 subjects.

SECONDARY OUTCOMES:
incidence of hepatotoxicity by genotypic variants | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deog Kyeom Kim, M.D., Study Director — SMG-SNUH Bormae Medical Center
Locations (1):
- Deog Kyeom Kim, Seoul, South Korea